CLINICAL TRIAL: NCT06731920
Title: The Incidence of Inadvertent Intravascular Injection During Ultrasound-guided Cervical Medial Branch Blocks: a Fluoroscopically Controlled Study
Brief Title: USG CMBB DSA Study
Status: Recruiting | Type: Observational
Sponsor: Montreal General Hospital (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Roderick Finlayson, RODERICK FINLAYSON MD, University of British Columbia
Other Study IDs: 2024-25-007-H
Record Dates: First submitted 2024-12-11; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Cervicalgia
Keywords: Ultrasound; cervical medial branch block; safety; digital subtraction angiography
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Main study group: Patients undergoing cervical medial branch blocks as part of their usual care.
  Interventions: Diagnostic Test: cervical medial branch block

INTERVENTIONS:
Diagnostic Test: cervical medial branch block — ultrasound-guided cervical medial branch block with fluoroscopic control and digital subtraction angiography

SUMMARY:
Injections that freeze neck joints can be done using x-rays or ultrasound imaging, which as a newer way of guiding the needle to the right spot. This study will look at how often freezing liquid goes into a blood vessel during neck injections that freeze neck joints when ultrasound guidance is used to place the needle. When this happens, it can go undetected because it does not make the patient feel any different, however it could cause a test block to be falsely negative, leading to the wrong diagnosis. Based on previous studies, we think that this happens rarely, and the purpose of this study is to prove that conclusively

DETAILED DESCRIPTION:
Cervical medial branch blocks (CMBB) are commonly employed for the diagnosis and management of facet-related pain. The latter constitutes the most important cause of axial neck pain and has been implicated in 40% of all cases. In addition, the upper cervical joints can also cause cervicogenic headaches, an often-debilitating condition representing up to 20% of chronic headaches3. Well-defined pain referral patterns for each joint can help operators select the appropriate injection level. While fluoroscopy has long been the imaging standard for spinal procedures, ultrasound guidance (USG) is being increasingly adopted as an alternative and presents several advantages such as the ability to identify and avoid soft tissue structures such as blood vessels during needle insertion. From a clinical perspective, avoiding blood vessels and reducing the incidence of vascular breach can lessen the occurrence of intravascular injections that are associated with false negative diagnostic blocks. Indeed, a recent study examining the safety of USG CMBB reported a lower incidence of vascular breach than previous studies that had used fluoroscopic guidance. While these findings suggested a potential benefit associated with USG, further confirmatory studies employing digital subtraction angiography (DSA), the current imaging standard to detect intravascular spread, are required. We hypothesize that USG will be associated will a lower incidence of intravascular spread during primary needle placement than has been reported with fluoroscopic guidance.

ELIGIBILITY:
Inclusion Criteria:

Consenting patients over 19 years of age undergoing an ultrasound-guided cervical medial branch blocks as part of their usual care.

Exclusion Criteria:

Subjects with one or more of the following characteristics will be excluded from the study:

Known bleeding disorder or coagulopathy Patients on antiplatelet medication other than aspirin and those on anticoagulants (coumadin, AT III agents) Inability to visualize targeted structures on ultrasound Known allergy to contrast agents

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cervical medial branch blocks as part of their usual care.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of vascular uptake | During the course of needle placement
  Incidence of intravascular spread of contrast as determined after a review of the DSA sequences by a physician not involved in the patient's care.

SECONDARY OUTCOMES:
Observed blood vessels | During needle placement
  Number and distribution of vessels observed near the target.
Incidence of vascular breach | During needle placement
  Incidence of vascular breach during needle placement.
Number of needle repositionings | During needle placement
  Number of needle repositionings required (before and after DSA)
Complications | From beginning to completion of block procedure
  Occurrence of any block-related complications.

CONTACTS AND LOCATIONS:
Overall Officials: Roderick J Finlayson, MD, Principal Investigator — University of British Columbia
Locations (1):
- Bill Nelems Pain and Research Centre, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No